CLINICAL TRIAL: NCT03472404
Title: Lateral Ligament Repair for Ankle Instability Protected With Internal Bracing. A Multicenter, Randomized Controlled Trial.
Brief Title: inStability Treated With Ligament RecOnstruction Augmented With iNternal bracinG
Acronym: STRONG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter van der Weegen (Other)
Collaborators: Medinova Clinics (Unknown); Gelre Hospitals (Other)
Responsible Party: Sponsor-Investigator, Walter van der Weegen, Principal Investigator, St. Anna Ziekenhuis, Geldrop, Netherlands
Organization: St. Anna Ziekenhuis, Geldrop, Netherlands (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W18.016
Record Dates: First submitted 2018-03-02; First posted 2018-03-21 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Ankle Sprains; Talofibular; Sprain (Strain)
MeSH Terms: conditions — Ankle Injuries; Sprains and Strains

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Internal Brace augmented ankle Ligament reconstruction
  Interventions: Procedure: Internal Brace augmented ankle Ligament reconstruction
- Control Group (Active Comparator): Brostrom-Gould ankle Ligament reconstruction
  Interventions: Procedure: Brostrom-Gould ankle Ligament reconstruction

INTERVENTIONS:
Procedure: Internal Brace augmented ankle Ligament reconstruction — internal brace augmented ankle ligament reconstruction and an accelerated revalidation protocol.
  Arms: Intervention Group
Procedure: Brostrom-Gould ankle Ligament reconstruction — Brostrom-Gould and standard revalidation including 6 weeks immobilisation.
  Arms: Control Group

SUMMARY:
This study evaluates the effect of internal bracing in lateral ligament ankle surgery. Half of the patients will receive the standard Brostrom-Gould reconstruction followed by a standard revalidation protocol including 6 weeks of immobilisation, while the other half of the patients will receive the same operation augmented with internal brace followed by an accelerated rehabilitation protocol.

DETAILED DESCRIPTION:
Ankle inversion trauma often leads to chronic ankle instability which can severely limit the patient during daily activities, including work and sports. When conservative treatment fails, surgical treatment in which the ruptured anterior talofibular ligament (ATFL) is reconstructed can be considered. Surgical treatment for ankle instability is associated with a relatively long rehabilitation due to the initial limited strength of the reconstructed ligament. This limited strength in the first weeks after surgery makes it necessary to protect the reconstructed lateral ankle ligament with immobilization. Usually a lower leg plaster is applied for six weeks. Due to the initial limited strength of the reconstructed ligament and the immobilization period itself, return to activities after surgery for this injury usually takes up to six months or even more. Therefore, surgical intervention is only indicated for patients who suffer chronic, recurrent ankle instability.

With a new surgical technique, an internal brace is placed over the reconstructed lateral ankle ligament, thereby providing protection which makes immobilization in the postoperative weeks unnecessary. This allows an earlier start of the rehabilitation which might enhance ankle function postoperatively and allows earlier return to activities. Also, adding an internal brace to the reconstructed lateral ankle ligament might result in a lower recurrence rate of ankle instability compared to the current surgical procedure.

Objective: To evaluate if patients with chronic, recurrent lateral ankle instability who are treated with surgical lateral ankle ligament repair protected with an internal brace, have significant better ankle function after surgery compared to patients treated with standard surgical lateral ankle ligament reconstruction without internal brace. The appropriately adapted rehabilitation for each surgery procedure is applied.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with chronic lateral ankle instability (multiple ankle inversion trauma within 12 months and symptoms present >1 year). Lateral ankle instability is present if the patient complains of giving way of the ankle and has positive signs of ankle instability during physical exam (talar tilt score of >15 degrees compared to contralateral ankle or anterior drawer test score of >10mm compared to the contralateral ankle.
* Conservative therapy has failed.
* Normal foot and ankle anatomy as determined by orthopedic surgeon.
* Patients in whom their ankle symptoms interfere with their physical activities.
* Patients with isolated anterior talofibular ligament which is indicated for repair using the Brostrom-Gould technique.
* BMI ≤30
* Patients who are able and willing to undergo ankle surgery.
* Patients who are able and willing to comply with the rehabilitation protocol in any of the study physiotherapy centers.
* Patients who are able and willing to return for follow-up evaluations.
* Patients with sufficient understanding of the Dutch language.

Exclusion Criteria:

* Patients who need concomitant ankle surgery (i.e. Calcaneofibular ligament reconstruction, peroneus tendon repair, arthroscopy of the ankle, etc).
* Patients with comorbidities, including musculoskeletal injuries or diseases in other joints than the affected ankle which limits their physical activity.
* Ankle instability due to abnormal foot and ankle anatomy.
* No objective or subjective ankle instability.
* Previous ankle surgery.
* Patients in which the contralateral ankle also shows lateral ankle instability.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Foot Ankle Outcome Score (FAOS) at 12 months | pre-operative, post-operative at 12 months
  Patient reported outcome measure, consists of 42 items, each item is scored in a 5-point likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Walter van der Weegen, Dr., Principal Investigator — St. Anna Hospital
Locations (3):
- Netherlands (3):
  - Gelre Ziekenhuis, Apeldoorn
  - Medinova, Breda
  - St Anna hospital, Geldrop

IPD SHARING:
Plan to Share IPD: No